CLINICAL TRIAL: NCT05313789
Title: Analgesia Nociception Index for Pain Monitoring in Intensive Care Units
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Principal Investigator, Ali Sefik Koprulu, MD, Ass. Prof., Ass. Prof., İstanbul Yeni Yüzyıl Üniversitesi
Other Study IDs: 20180413.2018/04-2
Record Dates: First submitted 2022-03-16; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Stress Related Disorder; Pain; Intensive Care Unit Syndrome
Keywords: Analgesia Nociception Index; Intensive Care Unit; Pain Monitoring
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intensive Care Patients (Cardiovascular): Intensive care unit patients, mechanically ventilated and lacking communication. Will examine whether the positive inotropic/vasoconstrictor agents will have any effect on Analgesia Nociception Index.
  Interventions: Device: Analgesia Nociception Index (ANI)
- Intensive Care Patients (Internal diseases): Intensive care unit patients, both mechanically ventilated and lacking communication and mechanically ventilated and conscious. Will examine whether the positive inotropic/vasoconstrictor agents will have any effect on Analgesia Nociception Index.
  Interventions: Device: Analgesia Nociception Index (ANI)
- Intensive Care Patients (Obese): Intensive care unit patients. Will examine whether the positive inotropic/vasoconstrictor agents will have any effect on Analgesia Nociception Index.
  Interventions: Device: Analgesia Nociception Index (ANI)

INTERVENTIONS:
Device: Analgesia Nociception Index (ANI) — Monitorization of Analgesia Nociception Index in Intensive Care Patients

SUMMARY:
The aim of this study is to examine the usability of ANI in patients who will be treated in intensive care unit.

DETAILED DESCRIPTION:
The aim of this study is to examine the usability of Analgesia Nociception Index in patients who will be treated in intensive care unit ( a- Cardiovascular b- surgical c- internal diseases), mechanically ventilated and lacking communication. The investigators will examine whether the positive inotropic/vasoconstrictor agents will have any effect on Analgesia Nociception Index.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care Cardiovascular Patients Group 1 - Patients aged from 18 to 80 years, scheduled for elective isolated coronary bypass graft (CABG) for 2-4 vessel disease, without any perioperative complications, and who were postoperatively monitored via the analgesia nociception index in the cardiovascular intensive care will be included.
* Intensive Care Internal Diseases Group 2 - Patients aged from 18 to 80 years, intubated or tracheostomized, In mechanical ventilation with Pressure-Controlled Ventilation mode, under perfusion neuromuscular blocker, Normothermic, non-cooperative and/or sedated and neuromuscular blocker
* Intensive Care Patients (Obese) Group 3 - Post Bariatric surgery, over 40 BMI

Exclusion Criteria:

* Intensive Care Cardiovascular Patients Group 1 Patients who required emergency surgery, had significant preoperative chronic pain, had autonomic nervous system anomalies and patients with rhythm will be excluded from the study.
* Intensive Care Internal Diseases Group 2 Ramsey sedation scale under 5, cooperative, with spontaneous breathing effort and extremity movement, non sinusal cardiac rhythm
* Intensive Care Patients (Obese) Group 3 - patients under 40 BMI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients between 18 and 80 years old. White Turkish Population.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-04-11 (Estimated); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
Analgesia Nociception Index for pain monitorization | 3 Months
  The duration between two R waves within heart rate variations (filtering the variations in respiratory cycles). A numeric measure of parasympathetic tonus will be obtained. This variation is between (pΣ) 0 and 100.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Guen M, Jeanne M, Sievert K, Al Moubarik M, Chazot T, Laloe PA, Dreyfus JF, Fischler M. The Analgesia Nociception Index: a pilot study to evaluation of a new pain parameter during labor. Int J Obstet Anesth. 2012 Apr;21(2):146-51. doi: 10.1016/j.ijoa.2012.01.001. Epub 2012 Feb 21. PMID 22360936
- [Background] Jeanne M, Clement C, De Jonckheere J, Logier R, Tavernier B. Variations of the analgesia nociception index during general anaesthesia for laparoscopic abdominal surgery. J Clin Monit Comput. 2012 Aug;26(4):289-94. doi: 10.1007/s10877-012-9354-0. Epub 2012 Mar 28. PMID 22454275
- [Background] Dias Dde S, Resende MV, Diniz Gdo C. Patient stress in intensive care: comparison between a coronary care unit and a general postoperative unit. Rev Bras Ter Intensiva. 2015 Jan-Mar;27(1):18-25. doi: 10.5935/0103-507X.20150005. Epub 2015 Mar 1. PMID 25909309
- [Background] Soral M, Altun GT, Dincer PC, Arslantas MK, Aykac Z. Effectiveness of the Analgesia Nociception Index Monitoring in Patients Who Undergo Colonoscopy with Sedo-Analgesia. Turk J Anaesthesiol Reanim. 2020 Feb;48(1):50-57. doi: 10.5152/TJAR.2019.45077. Epub 2019 Sep 24. PMID 32076680
- [Background] Jendoubi A, Abbes A, Ghedira S, Houissa M. Pain Measurement in Mechanically Ventilated Patients with Traumatic Brain Injury: Behavioral Pain Tools Versus Analgesia Nociception Index. Indian J Crit Care Med. 2017 Sep;21(9):585-588. doi: 10.4103/ijccm.IJCCM_419_16. PMID 28970658
- [Background] Broucqsault-Dedrie C, De Jonckheere J, Jeanne M, Nseir S. Measurement of Heart Rate Variability to Assess Pain in Sedated Critically Ill Patients: A Prospective Observational Study. PLoS One. 2016 Jan 25;11(1):e0147720. doi: 10.1371/journal.pone.0147720. eCollection 2016. PMID 26808971